CLINICAL TRIAL: NCT00052754
Title: Phase II Study Of Iressa (ZD 1839) In Locally Advanced And/Or Metastatic Synovial Sarcoma Expressing HER1/EGFR1
Brief Title: Gefitinib in Treating Patients With Locally Advanced or Metastatic Synovial Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62022; EORTC-62022
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Sarcoma
Keywords: adult synovial sarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Biological therapies such as gefitinib may interfere with the growth of the tumor cells and slow the growth of synovial sarcoma.

PURPOSE: Phase II trial to study the effectiveness of gefitinib in treating patients who have locally advanced or metastatic synovial sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic activity of gefitinib, in terms of progression-free rate, in patients with locally advanced or metastatic synovial sarcoma expressing HER1.
* Determine the toxicity of this drug in these patients.
* Determine the objective response, in terms of time to onset and duration of response, in patients treated with this drug.
* Determine the overall survival of patients treated with this drug.

OUTLINE: This is a non-randomized, multicenter study.

Patients receive oral gefitinib twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 14-44 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven advanced or metastatic synovial sarcoma that is not amenable to surgery, radiotherapy, or combined modality treatment with curative intent
* HER1 antigen expression
* Must have received at least 1 prior chemotherapy regimen comprising doxorubicin and/or ifosfamide
* At least 1 measurable lesion with evidence of progression within 3 months of study

  * Osseous lesions and pleural effusions are not considered measurable
* No symptomatic or known CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 3,000/mm^3
* Granulocyte count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Albumin at least 25 g/L

Renal

* Creatinine no greater than 2 times ULN OR
* Creatinine clearance greater than 65 mL/min

Cardiovascular

* No history of severe cardiovascular disease

Pulmonary

* No evidence of clinically active interstitial lung disease

  * Asymptomatic chronic stable radiographic changes allowed

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known severe hypersensitivity to gefitinib or any of its excipients
* No other primary malignant tumor except adequately treated carcinoma in situ of the cervix, basal cell skin cancer, or any other malignant tumor in complete remission for at least 3 years
* No other severe medical illness
* No psychosis
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 28 days since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 months since prior radiotherapy to measurable lesion and recovered
* No concurrent radiotherapy for soft tissue sarcoma
* Concurrent palliative radiotherapy to nontarget lesions allowed

Surgery

* Not specified

Other

* More than 28 days since prior unapproved or investigational drugs and recovered
* No concurrent phenytoin, carbamazepine, rifampin, barbiturates, or Hypericum perforatum (St. John's Wort)
* No other concurrent cytostatic agents
* No other concurrent tyrosine kinase activity inhibitors
* No other concurrent systemic therapy for soft tissue sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-10; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Progression-free rate at 12 weeks

SECONDARY OUTCOMES:
Toxicity as assessed by CTC 2.0
Response as assessed by RECIST criteria
Time to onset of response
Duration of response
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Blay, MD, PhD, Study Chair — Centre Leon Berard
Locations (16):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - U.Z. Gasthuisberg, Leuven
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie - Section Medicale, Paris
  - Institut Gustave Roussy, Villejuif
- Netherlands (4):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Leiden University Medical Center, Leiden
  - Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
- United Kingdom (4):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Marsden NHS Foundation Trust - London, London, England
  - Meyerstein Institute of Oncology at University College of London Hospitals, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England

REFERENCES:
- [Result] Ray-Coquard I, Le Cesne A, Whelan JS, Schoffski P, Bui BN, Verweij J, Marreaud S, van Glabbeke M, Hogendoorn P, Blay JY. A phase II study of gefitinib for patients with advanced HER-1 expressing synovial sarcoma refractory to doxorubicin-containing regimens. Oncologist. 2008 Apr;13(4):467-73. doi: 10.1634/theoncologist.2008-0065. PMID 18448563